CLINICAL TRIAL: NCT03502746
Title: Phase II Study of Nivolumab and Ramucirumab for Patients With Previously-Treated Mesothelioma:Hoosier Cancer Research Network LUN15-299
Brief Title: Phase II Nivolumab and Ramucirumab for Patients With Previously-Treated Mesothelioma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: IRB Study Closure
Sponsor: Arkadiusz Z. Dudek, MD (Other)
Collaborators: HealthPartners Institute Regions Cancer Care Center (Other); Eli Lilly and Company (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Arkadiusz Z. Dudek, MD, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCRN-LUN15-299
Record Dates: First submitted 2018-04-11; First posted 2018-04-19 (Actual); Results first posted 2023-10-26 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-04

CONDITIONS: Mesothelioma, Malignant
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Nivolumab; Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab + Ramucirumab (Experimental): Nivolumab 240mg IV + Ramucirumab 8mg/kg IV
  Interventions: Drug: Nivolumab; Drug: Ramucirumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 240mg, IV over 30 minutes.
  Other Names: Opdivo
Drug: Ramucirumab — 8mg/kg, IV over 60 minutes.
  Other Names: Cyramza

SUMMARY:
This study will evaluate the combination of Nivolumab and Ramucirumab in patients with previously-treated mesothelioma.

DETAILED DESCRIPTION:
The programmed death ligand 1 (PD-L1) [16] and VEGFR2 [34] are highly-expressed on mesothelioma cells, and are therefore attractive options for this cancer. We chose to study the combination of ramucirumab with nivolumab because of the potential efficacy of these two agents in mesothelioma and because of the potential synergistic activity between them [30]. As previously discussed, immunotherapies such as anti-PD-1 inhibitors must contend with a hostile, immunosuppressive tumor microenvironment due to angiogenesis that results in hypoxia. This hypoxia decreases the ability of antibodies to infiltrate the tumor. We hypothesize that the normalization of tumor vasculature (by reducing the area of the tumor that is hypoxic) with an anti-VEGF strategy (i.e., ramucirumab) used in synergy with a PD-1 inhibitor will facilitate the infiltration of T-lymphocytes into tumor parenchyma. We will conduct a phase II study based on this premise using nivolumab and ramucirumab as second-line therapy in patients with malignant mesothelioma who have failed standard doublet platinum and anti-folate therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age at time of consent.
* Histologically-confirmed malignant mesothelioma not amenable to curative surgery and who have received at least one pemetrexed-containing chemotherapy regimen.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* total bilirubin < 1.5 mg/dL (25.65 μmol/L) OR direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 mg/dL (except subject with Gilbert's Syndrome, who can have total bilirubin < 3.0 mg/dl)
* aspartate aminotransferase (AST) ≤ 3 × ULN or ≤ 5 × ULN for subjects with known hepatic metastases
* alanine aminotransferase (ALT) ≤ 3 × ULN or ≤ 5 × ULN for subjects with known hepatic metastases
* hemoglobin ≥ 8 g/dL, subjects requiring transfusion will not be eligible to start study
* absolute neutrophil count (ANC) ≥ 1.5 × 109/L
* platelet count ≥ 100 × 109/L
* serum creatinine ≤1.5 times the ULN, or creatinine clearance (measured via 24-hour urine collection) ≥40 mL/minute (that is, if serum creatinine is >1.5 times the ULN, a 24-hour urine collection to calculate creatinine clearance must be performed)
* subject's urinary protein is ≤1+ on dipstick or routine urinalysis (UA; if urine dipstick or routine analysis is ≥2+, a 24-hour urine collection for protein must demonstrate <1000 mg of protein in 24 hours to allow participation in this protocol)
* INR < 1.5, and a partial thromboplastin time (PTT) (PTT/aPTT) < 1.5 x ULN (unless receiving anticoagulant therapy)
* Subjects on full-dose anticoagulation must be on a stable dose (minimum duration 14 days) of oral anticoagulant or low molecular weight heparin (LMWH). Patients receiving warfarin must be switched to low molecular weight heparin and have achieved stable coagulation profile prior to first dose of protocol therapy. For heparin and LMWH there should be no active bleeding (that is, no bleeding within 14 days prior to first dose of protocol therapy) or pathological condition present that carries a high risk of bleeding (for example, tumor involving major vessels or known varices).
* Subjects must be willing to undergo a CT-guided biopsy (i.e., image-guided percutaneous lung biopsy) to obtain tumor tissue within 28 days before initiation of treatment and after 4 cycles (8 weeks) of treatment.
* Women of childbearing potential (WOCP) must be willing to use birth control as outlined in the protocol.
* Men who are not surgically or medically sterile must agree to use contraception as outlined in the protocol.
* Measurable disease, defined as at least 1 tumor that fulfills the criteria for a target lesion according to modified RECIST 1.1 criteria, and obtained by imaging within 28 days prior to study registration.
* Prior intracavity cytotoxic or sclerosing agents (including bleomycin) is acceptable.
* Radiation therapy must be completed > 28 days before study registration, and the measurable disease must be outside of the radiation port.
* Pemetrexed-containing chemotherapy must be completed > 28 days before study registration.
* Must provide written informed consent and HIPAA authorization approved by an Institutional Review Board (IRB). NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* All previous toxicity resolved to Grade 1 or less.

Exclusion Criteria:

* Any Grade 3-4 GI bleeding within 3 months prior to study registration.
* History of deep vein thrombosis, pulmonary embolism, or any other significant thromboembolism (venous port or catheter thrombosis or superficial venous thrombosis are not considered "significant") during the 3 months prior to study registration.
* Any arterial thromboembolic events, including but not limited to myocardial infarction, transient ischemic attack, cerebrovascular accident, or unstable angina, within 6 months prior to study registration.
* Cirrhosis at a level of Child-Pugh B (or worse), or cirrhosis (any degree) with a history of hepatic encephalopathy, or clinically meaningful ascites resulting from cirrhosis. Clinically meaningful ascites is defined as ascites from cirrhosis requiring diuretics or paracentesis.
* Uncontrolled or poorly-controlled hypertension (>160 mmHg systolic or > 100 mmHg diastolic for >4 weeks) despite standard medical management.
* Prior history of GI perforation/fistula (within 6 months of study registration) or risk factors for perforation.
* Serious or nonhealing wound, ulcer, or bone fracture within 28 days prior to study registration.
* Active brain metastases or carcinomatous meningitis. Subjects with neurological symptoms must undergo a head CT scan or brain MRI to exclude brain metastasis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of study drugs and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 14 days prior to study registration. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability.
* Major surgery within 28 days prior to study registration
* Subcutaneous venous access device placement within 7 days prior to study registration.
* Elective or planned major surgery to be performed during the course of the clinical trial.
* Is receiving chronic antiplatelet therapy, including aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs, including ibuprofen, naproxen, and others), dipyridamole or clopidogrel, or similar agents. Once-daily aspirin use (maximum dose 325 mg/day) is permitted.
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS). NOTE: HIV testing is not required.
* Known history of testing positive for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody), indicating acute or chronic infection. NOTE: Hepatitis B and Hepatitis C testing is not required.
* Condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.

  o NOTE: Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Received a live vaccine within 30 days prior to the first dose of trial treatment. Examples of live vaccines include, but are not limited to: measles, mumps, rubella, chicken pox, yellow fever, rabies, BCG, and typhoid (oral) vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g. Flu-Mist®) are live attenuated vaccines and are not allowed.
* History of interstitial lung disease or active, non-infectious pneumonitis.
* Female subject is pregnant or breast-feeding.

  * NOTE: Women of childbearing potential (WOCP) must have a negative pregnancy test (either serum β-HCG with a sensitivity of 50 mIU/ml or urine dipstick within 24 hours of study registration).
  * NOTE: Women are not considered to be of childbearing potential if they meet at least one of the following: 1) surgically sterilized, or 2) postmenopausal (a woman who is ≥45 years of age and has not had menses for greater than 1 year), or 3) not heterosexually active for the duration of the study. See section 5.6.2.
* Major blood vessel invasion or significant intratumor cavitation.
* If they experience hemoptysis (defined as bright red blood or ≥ ½ teaspoon) within 2 months prior to first dose of protocol therapy or with radiographic evidence of intratumor cavitation or has radiologically documented evidence of major blood vessel invasion or encasement by cancer.
* Any condition that, in the opinion of the investigator, might jeopardize the safety of the subject or interfere with protocol compliance.
* Any mental or medical condition that prevents the subject from giving informed consent or participating in the trial.
* Any pathological condition that carries a high risk of bleeding (for example, tumor involving major vessels or known varices.)
* Known hypersensitivity to nivolumab or ramucirumab or any of their components.
* Known history of active tuberculosis.
* Received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* No prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, localized Gleason ≤ grade 7 prostate cancers. Subjects with other solid tumors treated curatively and without evidence of recurrence for at least 3 years prior to enrollment may be eligible for study after discussion with the sponsor-investigator
* Treatment with any investigational agent within 28 days prior to study registration. The subject must have recovered from the acute toxic effects of the regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2023-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arkadiusz Z Dudek, MD, Principal Investigator — HealthPartners Institute Regions Cancer Care Center
Locations (4):
- United States (4):
  - Moffitt Cancer Center, Tampa, Florida
  - University of Maryland, Baltimore, Maryland
  - Karmanos Cancer Center (Wayne State University), Detroit, Michigan
  - HealthPartners Institute Regions Cancer Care Center, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dudek AZ, Xi MX, Scilla KA, Mamdani H, Creelan BC, Saltos A, Tanvetyanon T, Chiappori A. Phase 2 Trial of Nivolumab and Ramucirumab for Relapsed Mesothelioma: HCRN-LUN15-299. JTO Clin Res Rep. 2023 Oct 12;4(12):100584. doi: 10.1016/j.jtocrr.2023.100584. eCollection 2023 Dec. PMID 38046376

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nivolumab + Ramucirumab
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Nivolumab + Ramucirumab
Number analyzed (Participants) | 34
Age, Continuous [Median (Full Range); unit: years] | 72 [40 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 31
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34
Histology [Count of Participants; unit: Participants] — The pleura is the serous membrane which forms the lining of the pleural cavity and the peritoneum is the serous membrane covering the abdominal cavity.
  Participants
    Pleural | 30
    Peritoneal | 4

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD. Response rate will be defined as the proportion of all subjects with confirmed PR or CR according to RECIST 1.1.
Time Frame: Up to a maximum of 23 months
Population: Out of 34 patients, one patient was not evaluable for response after he withdrew from study because of generalized weakness one day after first infusion of ramucirumab and nivolumab.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab + Ramucirumab
Number analyzed (Participants) | 33
Percentage of participants | 22.6 [9.6 to 41.1]

2. Secondary Outcome: Adverse Event Assessment
Description: The frequency and severity of all grade ≥ 2 treatment related adverse events are reported by CTCAE v4 term.
Time Frame: AE had been recorded from time of consent until 100 days after discontinuation of study drug or until a new anti-cancer treatment starts, whichever occurs first; up to a maximum of 28 months.
Measure: Number; unit: Participants
Arm/Group | Nivolumab + Ramucirumab
Number analyzed (Participants) | 34
Participants
  Dyspnea | 5
  Hypertension | 3
  Proteinuria | 9
  Arial fibrillation | 2
  Abdominal Pain | 1
  Anorexia | 2
  Dehydration | 1
  Diarrhea | 1
  Dysphagia | 1
  Esophageal Obstruction | 1
  Fatigue | 7
  Hyperkalemia | 1
  Hyponatremia | 1
  Muscle Weakness | 3
  Non-Cardiac Chest Pain | 1
  Pancreatitis | 1
  Thromboembolic Event | 1
  Pain | 3
  Sinusitis | 3
  Depression | 2
  Hypothyroidism | 2
  Dizziness | 2
  Chest Wall Pain | 1
  Cough | 1
  Creatinine Increased | 1
  Heart Failure | 1
  Hypoxia | 1
  Lower Gastrointestinal Bleed | 1
  Mucositis Oral | 1
  Periodontal Disease | 1
  Pneumonitis | 1
  Presyncope | 1
  Weight loss | 1
  Atopic Dermatitis | 1
  Upper Respiratory Tract Infection | 1

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD. PFS is defined as time from treatment start until disease progression met by RECIST 1.1 or death from any cause.
Time Frame: Time of treatment start until the criteria for disease progression or death, up to a maximum of 23 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab + Ramucirumab
Number analyzed (Participants) | 34
Months | 4.2 [1.9 to 6.4]

4. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined as time of treatment start until death or date of last contact.
Time Frame: Time of treatment start until death or date of last contact, up to a maximum of 32 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab + Ramucirumab
Number analyzed (Participants) | 34
Months | 12.5 [6.3 to 23.5]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored up to a maximum of 32 months. Serious Adverse Events and Other (Not Including Serious) Adverse Events were monitored up to 28 months.
Arm/Group | Nivolumab + Ramucirumab
All-Cause Mortality (participants affected / at risk) | 22/34
Serious Adverse Events (participants affected / at risk) | 9/34
Other Adverse Events (participants affected / at risk) | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab + Ramucirumab (N=34)
ATRIAL FIBRILLATION (Cardiac disorders) | 2 (2)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ESOPHAGEAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1)
HEART FAILURE (Cardiac disorders) | 1 (1)
LOWER GASTROINTESTINAL HEMORRHAGE (Gastrointestinal disorders) | 1 (1)
MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab + Ramucirumab (N=34)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 2 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1)
ALLERGIC REACTION (Immune system disorders) | 1 (1)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ANEMIA (Blood and lymphatic system disorders) | 1 (3)
ANOREXIA (Metabolism and nutrition disorders) | 10 (12)
ANXIETY (Psychiatric disorders) | 2 (3)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5 (5)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 3 (3)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 (5)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
CHEST WALL PAIN (Musculoskeletal and connective tissue disorders) | 4 (5)
CHILLS (General disorders) | 2 (2)
CONFUSION (Psychiatric disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 3 (3)
COUGH (Respiratory, thoracic and mediastinal disorders) | 11 (12)
CREATININE INCREASED (Investigations) | 3 (6)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1)
DEPRESSION (Psychiatric disorders) | 3 (3)
DIARRHEA (Gastrointestinal disorders) | 5 (9)
DIZZINESS (Nervous system disorders) | 4 (4)
DRY SKIN (Skin and subcutaneous tissue disorders) | 4 (4)
DYSGEUSIA (Nervous system disorders) | 2 (2)
DYSPHAGIA (Gastrointestinal disorders) | 1 (2)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 7 (11)
EDEMA LIMBS (General disorders) | 7 (8)
EDEMA TRUNK (General disorders) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (2)
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 3 (3)
FATIGUE (General disorders) | 19 (22)
FEVER (General disorders) | 1 (1)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - OTHER, SPECIFY (General disorders) | 3 (4)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 7 (7)
GLUCOSE INTOLERANCE (Metabolism and nutrition disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 6 (10)
HEMATURIA (Renal and urinary disorders) | 2 (2)
HEMORRHOIDS (Gastrointestinal disorders) | 2 (2)
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 2 (4)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 (1)
HYPERKALEMIA (Metabolism and nutrition disorders) | 1 (9)
HYPERMAGNESEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPERTENSION (Vascular disorders) | 3 (6)
HYPERTHYROIDISM (Endocrine disorders) | 1 (1)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOKALEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 3 (5)
HYPONATREMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOTHYROIDISM (Endocrine disorders) | 4 (6)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 1 (1)
INFUSION RELATED REACTION (General disorders) | 3 (5)
INFUSION SITE EXTRAVASATION (General disorders) | 1 (3)
INSOMNIA (Psychiatric disorders) | 1 (1)
IRRITABILITY (General disorders) | 1 (2)
MEMORY IMPAIRMENT (Nervous system disorders) | 2 (2)
MUCOSITIS ORAL (Gastrointestinal disorders) | 2 (2)
MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCLE WEAKNESS UPPER LIMB (Musculoskeletal and connective tissue disorders) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 4 (5)
NAUSEA (Gastrointestinal disorders) | 6 (6)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2)
NON-CARDIAC CHEST PAIN (General disorders) | 4 (4)
PAIN (General disorders) | 10 (13)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 (4)
PAROXYSMAL ATRIAL TACHYCARDIA (Cardiac disorders) | 1 (1)
PERIODONTAL DISEASE (Gastrointestinal disorders) | 1 (1)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 2 (2)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PRESYNCOPE (Nervous system disorders) | 1 (1)
PROTEINURIA (Renal and urinary disorders) | 9 (25)
PRURITUS (Skin and subcutaneous tissue disorders) | 2 (3)
PURPURA (Skin and subcutaneous tissue disorders) | 1 (1)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 5 (5)
RENAL AND URINARY DISORDERS - OTHER, SPECIFY (Renal and urinary disorders) | 1 (1)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (Respiratory, thoracic and mediastinal disorders) | 1 (2)
SINUS TACHYCARDIA (Cardiac disorders) | 1 (2)
SINUSITIS (Infections and infestations) | 1 (1)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (Skin and subcutaneous tissue disorders) | 4 (5)
SKIN HYPOPIGMENTATION (Skin and subcutaneous tissue disorders) | 1 (1)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 2 (2)
STOMACH PAIN (Gastrointestinal disorders) | 5 (5)
THROMBOEMBOLIC EVENT (Vascular disorders) | 1 (1)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 1 (2)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 2 (2)
VOMITING (Gastrointestinal disorders) | 3 (3)
WATERING EYES (Eye disorders) | 1 (1)
WEIGHT LOSS (Investigations) | 5 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/46/NCT03502746/Prot_SAP_000.pdf